CLINICAL TRIAL: NCT07055945
Title: Investigation of the Effects of Visual-Motor Based Training on Upper Extremity Functions in Individuals With Stroke
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Baskent University (Other)
Collaborators: Baskent University Ankara Hospital (Other)
Responsible Party: Principal Investigator, Ayşegül Aykul, Principal Investigator, MSc, Baskent University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: BUAYKUL-001
Record Dates: First submitted 2025-05-07; First posted 2025-07-09 (Actual); Last update posted 2025-09-04 (Actual); Status verified 2025-08

CONDITIONS: Stroke
Keywords: Stroke; Physiotherapy Rehabilitation; Functionality
MeSH Terms: conditions — Stroke | interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: The study consists of two groups: the visual-motor based training and physiotherapy program group and the physiotherapy program group. Both groups will receive a physiotherapy program for 60 minutes of 3 sessions per week for a total of 8 weeks. Patients from both groups will take 30 minutes of functional exercises. These exercises are fundamental and will be tailored to the individual needs of the patient. Light Trainer will be used for visual-motor based training in the experimental group.
Who Masked: Participant
Masking Description: A single-blind study was designed in which the patients would be unaware of their group allocation
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Visual-motor based training and physiotherapy program (Experimental): The physiotherapy group will take a physiotherapy program for 3 sessions per week, 60 minutes per day, for a total of 8 weeks. The program will consist of functional exercises for trunk, upper and lower extremities.
  In addition to the functional exercises individuals will receive visual-motor training targeting the upper extremity. This training will be conducted using the Light Trainer, a branded light-based training system. The light training system consists of 6 laser sensor-equipped blue, red, and green light emitters.The system is operated through a smartphone application.The training will utilize four different games, progressing from easy to difficult: Sequential, random standard, multiple light, and different color. Participants will receive training via a 12-minute session utilizing the Light Trainer device.
  Interventions: Other: Experimental group
- Physiotherapy group (Active Comparator): The physiotherapy group will take a physiotherapy program for 3 sessions per week, 60 minutes per day, for a total of 8 weeks.
  The program will consist of functional exercises for trunk, upper and lower extremities (same as experimental group).
  Functional reaching activities at the table in a sitting position, ball sliding on the wall in a standing position, touching different targets on the wall in a standing position and drawing shapes on the wall in a standing position will also added to the program.
  Interventions: Other: Control group

INTERVENTIONS:
Other: Experimental group — Individuals in both groups will receive a physiotherapy program for 3 sessions per week, 60 minutes per day, for a total of 8 weeks.The study consists of two groups: the experimental group and the control group. Both groups will receive a physiotherapy program of 3 sessions per week, each lasting 60 minutes, for a total of 8 weeks. Within the 60-minute physiotherapy session, patients from both groups will undergo 30 minutes of exercises based on the Neurodevelopmental Treatment (NDT) method. In addition, a 12-minute training session will be conducted using a light-based trainer system (Light Trainer® Exercise System).
  Arms: Visual-motor based training and physiotherapy program
Other: Control group — In addition to the full-body exercises mentioned, individuals in the control group will also receive upper extremity exercises based on the Neurodevelopmental Treatment approach. These exercises are as follows:
  * Functional reaching activities at the table in a sitting position (e.g., pushing objects, wiping the table, touching various points)
  * Ball sliding on the wall in a standing position
  * Touching different targets on the wall in a standing position
  * Drawing shapes on the wall in a standing position
  These exercises will be performed bilaterally and on the hemiparetic side. The exercises will be given for approximately 12 minutes, in line with the exercises given to the experimental group. The difficulty level will not be increased during the training.
  Arms: Physiotherapy group

SUMMARY:
The purpose of this study is to investigate the effects of visual-motor based training and physiotherapy program on upper extremity functions in individuals with stroke and to compare with physiotherapy program.

DETAILED DESCRIPTION:
Stroke is a clinical syndrome characterized by the sudden onset of signs and symptoms due to a localized loss of cerebral function, in the absence of any apparent cause other than a vascular origin.More than 50% of patients experience various impairments and dependence on others following a stroke. One of the primary reasons for this condition is problems affecting the upper extremity.

The Light Trainer system allows for the repetitive and non-repetitive practice of an activity. It enables goal-oriented, active participation, providing an enjoyable experience that engages the whole body. The difficulty level can be adjusted and is tailored to the individual's response ability. With these features, it supports motor learning. Given these characteristics, the Light Trainer system is considered suitable for use in patients with sensory-motor-cognitive disorders, such as those with stroke, multiple sclerosis, and Parkinson's disease. A literature review reveals that task-oriented exercises and virtual reality are commonly used for visual-motor training; however, no studies have been found involving this new system

The first aim of this study is to investigate the effects of visual-motor based training and physiotherapy program on upper extremity functions in individuals with stroke and to compare with physiotherapy program.

The second aim of this study is to investigate the effects of visual-motor based training and physiotherapy program on cognitive functions and trunk in individuals with stroke and to compare with physiotherapy program.

ELIGIBILITY:
Inclusion criteria:

* At least 6 months have passed since the cerebrovascular event
* Aged between 18 and 75 years
* First-time stroke
* Scoring 24 or higher on the Standardized Mini Mental Test (SMMT)
* Upper extremity functioning at Stage 4 or above according to the Brunnstrom Staging
* Shoulder, elbow, wrist, and finger muscle tone at or below a score of 2 on the Modified ---Ashworth Scale (MAS)
* Shoulder joint range of motion of at least 120°
* Ability to stand independently

Exclusion Criteria:

* Presence of hemispatial neglect syndrome
* Ataxia due to posterior circulatory ischemia
* Bilateral involvement (bilateral hemiparesis)
* Botulinum toxin injection in the last three months
* Physiotherapy treatment within the last 6 months
* Orthopedic problems such as shoulder subluxation, shoulder pain, or contractures in the hand or wrist
* Previous upper extremity or thoracic surgery
* Vision problems related to stroke (hemianopsia)
* Color blindness

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2025-08-28 (Actual); Primary Completion 2025-12-15 (Estimated); Study Completion 2025-12-30 (Estimated)

PRIMARY OUTCOMES:
Modified Ashworth Scale | eight weeks
  Modified Ashworth Scale (MAS) will be used to evaluate the muscle tone of the **shoulder, elbow, wrist, and finger flexors** in post-stroke patients. This scale will be applied both as part of the **initial assessment** for determining eligibility and to evaluate the **effectiveness of the intervention** by comparing pre- and post-treatment scores. MAS grades muscle tone on a 6-point ordinal scale.Each measurement will be performed twice. Data will be entered into the statistical database both as ordinal values (0 to 4) and using a coding system for further analysis. Patients will be evaluated pre- and post-treatment using the MAS.
Fugl-Meyer Upper Extremity Assessment | eight weeks
  The Fugl-Meyer Motor Assessment Scale is a performance-based motor impairment scale developed to evaluate recovery in individuals with stroke. This scale includes subtests that assess upper and lower extremity functions, balance, sensation, and posture. In our study, the upper extremity gross and fine motor functions of patients will be assessed using the Fugl-Meyer Upper Extremity (FM-UE) Assessment Scale. The maximum score that can be obtained in the assessment is 66, with higher scores indicating better motor function. Patients will be evaluated pre- and post-treatment using the Fugl-Meyer Assessment Scale.
Wolf Motor Function Test | eight weeks
  The Wolf Motor Function Test (WMFT) is a test developed to evaluate motor skills in patients with moderate to severe upper extremity motor deficits The original version was developed by Wolf and colleagues. In our study, the modified version developed by Morris and colleagues will be used.Data will be collected for 15 activities in two areas: "functional ability" and "performance time". The duration of the test is 30-45 minutes.Each activity will be rated by the physiotherapist using a scale of 0 to 5 based on the functional ability section, where:0 = "The affected hand is not used at all during the activity",5 = "Normal movement".The average score for functional ability will be calculated, and based on this, the patient will receive a score between 0 and 5, with higher scores indicating good functional ability.The performance time will be recorded in seconds.The maximum time given to complete an activity is 120seconds.Patients will be evaluated pre- and post-treatment using the WMFT
Purdue Pegboard Test | eight weeks
  The Purdue Pegboard Test(PPT) is used to assess the motor skills and coordination of the upper extremity. The test consists of a board with two parallel rows of 25 holes, along with pegs, rings, and small pins.In our study, upper extremity motor skills and coordination will be evaluated using the PPT. Scoring: Each pin inserted with the right or left hand earns 1 point, each pair of pins inserted with both hands earns 1 point, and each completed combination (pin, washer, and nut) is worth 4 points. Patients will be evaluated pre- and post-treatment using the PPT.

SECONDARY OUTCOMES:
Cognitive functions: Stroop Test-Interference Form | eight weeks
  The Stroop test is a cognitive assessment that evaluates executive functions and measures attention, the inhibition of inappropriate automatic responses, and perception under disruptive influence. The Stroop effect not only measures executive functions but also assesses processing speed, automatic, and parallel processing. The Stroop effect occurs when there is a conflict between the color name written and the color used to write it. When the colors are different, reading the word becomes slower compared to reading words that are written in the same color, and the difference between these two speeds is referred to as the Stroop effect. The Stroop effect not only measures executive functions but also assesses processing speed, automatic, and parallel processing. A longer completion time and a higher error count indicate weak cognitive flexibility. Patients will be evaluated pre- and post-treatment using the Stroop test.
Postural Assessment Scale for Stroke Patients | eight weeks
  The Postural Assessment Scale for Stroke Patients (PASS) is designed to evaluate postural control and balance in detail. The scale assesses balance during tasks such as lying, sitting, standing, or changing positions. Each task is rated from 0 (lowest) to 3 (highest). The total score ranges from 0 to 36. Higher scores on the PASS indicate better postural stability and functional independence, with a maximum score of 36 representing full postural competence. Patients will be evaluated pre- and post-treatment using the PASS.
Trunk functions: Body Disorder Scale (BDS) | eight weeks
  BDS is a tool used to assess motor dysfunctions resulting from stroke and to measure the quality of body movements. The scale consists of 17 parameters and is used to evaluate somatic, motor, and coordination deficits in stroke patients. The scale is divided into three subcategories: static sitting balance, dynamic sitting balance, and coordination. The total score ranges from 0 to 23 points, with higher scores indicating better performance. Patients will be evaluated pre- and post-treatment using the BDS.

CONTACTS AND LOCATIONS:
Overall Officials: Sevgi İkbali Afşar, Prof Dr, Study Director — Baskent University
Locations (1):
- Başkent University, Ankara, Türkiye, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
No, because all patient data are subject to the Başkent Hospital's patient privacy policy.